CLINICAL TRIAL: NCT01789450
Title: Nipple-Areola Complex Sensitivity After the Section of Periareolar Dermis in Breast Reduction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Jairo Zacchê de Sá, Jairo Zacchê de Sá, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UFPE
Record Dates: First submitted 2013-02-04; First posted 2013-02-12 (Estimated); Last update posted 2013-04-29 (Estimated); Status verified 2013-04

CONDITIONS: Sensitivity of Nipple-areolar Complex
Keywords: sensitivity; section of periareolar dermis; breast reduction
MeSH Terms: conditions — Hypersensitivity | interventions — Sensitivity and Specificity; Cerebral Decortication

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Section of Periareolar Dermis (Experimental): Section of Periareolar Dermis
  Interventions: Procedure: Section of Periareolar Dermis in Breast Reduction.

INTERVENTIONS:
Procedure: Section of Periareolar Dermis in Breast Reduction.
  Other Names: Sensitivity; Nipple-Areolar Complex (NAC); Breast Reduction; Schwartzmann's Maneuver; Decortication

SUMMARY:
The purpose of this study is to evaluate the feasibility and sensitivity of nipple-areolar complex (NAC) prospectively due to the section of the dermis after decortication (Schwartzmann's maneuver), in 50 patients undergoing breast reduction surgery.

DETAILED DESCRIPTION:
Preservation of the dermis after decortication regions of the areola and periareolar is considered relevant by most plastic surgeons.

In patients whose CAP should be mobilized through large distances in order to correct breast ptosis, or in cases of dense breasts where noted little slip of skin over the breast parenchyma, the periareolar dermis causes limitation on the mobility of the NAC.

In clinical practice, there is a greater mobilization of NAC when making a careful section of the dermis after decortication. In contrast, the appearance of partial necrosis in these cases has become a rarity, as no case of total necrosis was observed.

Given the technical benefit observed due to greater mobilization, there is no report in the literature about how behaves the sensitivity of the NAC in these cases.

To evaluate the sensitivity of the NAC will be used Semmes-Weisnstein's monofilament. Each point will be obtained five measurements. The largest will be scorned and the lowest value. The final value of each point corresponds to an arithmetic mean of the three remaining values.

ELIGIBILITY:
Inclusion Criteria:

* Patients who willingly seek the service requesting breast reduction or mastopexy;
* Patients who after consultation with the surgeon who led the research presents realistic expectation, being safe with the possible outcome of the surgery;
* Patients who undertake to comply with the protocol previously presented and discussed with them;

Exclusion Criteria:

* Patients with prior breast surgery;
* Patients with body mass index (BMI) greater than 34.9;
* Patients with severe anemia;
* Patients with neurological disease;
* Patients with impairment cardiovascular;
* Metabolic diseases - diabetes;
* Patients with autoimmune disease;
* Menopausal patients
* Patients with collagen disease;
* Patients with psychiatric disorders.

Ages: 21 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2013-06; Primary Completion 2014-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Nipple-Areola Complex (NAC) Sensitivity | 3 weeks
  To evaluate the sensitivity of the NAC in breast reduction

SECONDARY OUTCOMES:
Nipple-Areola Complex (NAC) sensitivity | 6 weeks
  To evaluate the sensitivity of the NAC in breast reduction

OTHER OUTCOMES:
Nipple-Areola Complex sensitivity | 12 months
  To evaluate the sensitivity of the NAC in breast reduction

CONTACTS AND LOCATIONS:
Overall Officials: Jairo Z Sá, surgeon, Principal Investigator — Hospital das Clínicas da Universidade Federal de Pernambuco
Locations (1):
- Hospital das clínicas da UFPE, Recife, Pernambuco, Brazil